CLINICAL TRIAL: NCT02004977
Title: Improving High School Breakfast Environments
Acronym: breakFAST!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1111S06384; 1R01HL113235 (NIH)
Record Dates: First submitted 2013-11-12; First posted 2013-12-09 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm (Experimental): The role of the intervention arm (schools) is to improve access to the school breakfast program
  Interventions: Behavioral: Improve access to the school breakfast program
- Comparison arm (No Intervention): the role of the comparison arm (schools) is to maintain usual breakfast program at school

INTERVENTIONS:
Behavioral: Improve access to the school breakfast program — Access to the school breakfast program is defined as implementation of a grab-n-go cart outside of the school cafeteria, policy change allowing students to eat in the hallway and marketing of the program. in rural high schools.
  Other Names: improve access to school breakfast
  Arms: Intervention arm

SUMMARY:
The goals of this intervention study are to implement best practice strategies to expand and promote the school breakfast program and test the impact upon student participation rates among a) all 10th and 11th grade students and among a randomly selected cohort of 800 students b) total diet and body mass index and percent body fat inin 16 rural Minnesota school districts.

School-wide Primary Aim: Improve participation in the school breakfast program among high school students. Hypothesis: School-wide school breakfast program participation will be higher in the intervention versus comparison group.

DETAILED DESCRIPTION:
We will accomplish the following secondary aims using a random subsample of 800 incoming 10th and11th grade students.

Student-level Secondary Aims Secondary Aim 1: High school students in the intervention condition will decrease their rate of weight gain relative to height gain as measured by change in body mass index and percent body fat compared to students in the control condition. Hypothesis: Body mass index and percent body fat will be maintained or reduced in the treatment versus control group.

Secondary Aim 2: High school students in the intervention condition will maintain or decrease their energy intake while improving dietary intakes of low fat dairy, whole grains and fresh fruits compared to the control students.

Hypothesis: Energy intake (measured by 3, 24-hour recalls) will be maintained or reduced and intakes of low fat dairy, whole grains and fresh fruits will increase more in the intervention groups.

Secondary Aim 3: Compared to students in the control condition, high school students in the intervention condition will report receiving more support to eat school breakfast. Support will be social (increased peer and school support) or related to the school environment (satisfaction with serving locations and times, eating locations, foods and increased availability of low fat dairy, fruits and whole grains for breakfast).

Hypothesis: The treatment group will report receiving more social and school environment support for eating school breakfast than the comparison group (measured by a student survey).

ELIGIBILITY:
Inclusion Criteria:

Must be in 10th or 11th grade in school year 2013-14 Must have access to the internet Must have access to a phone

Exclusion Criteria for the Cohort:

Unable to read English Unable to speak English Pregnant Plan to move out of the school district within school year Not in school most mornings Eat breakfast 4 or more days a week

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 904 (Actual)
Dates: Start 2013-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn S Nanney, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Nanney MS, Leduc R, Hearst M, Shanafelt A, Wang Q, Schroeder M, Grannon KY, Kubik MY, Caspi C, Harnack LJ. A Group Randomized Intervention Trial Increases Participation in the School Breakfast Program in 16 Rural High Schools in Minnesota. J Acad Nutr Diet. 2019 Jun;119(6):915-922. doi: 10.1016/j.jand.2018.12.007. Epub 2019 Feb 14. PMID 30772298

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Comparison Arm
Started | 463 | 441
Completed | 409 | 436
Not Completed | 54 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Comparison Arm | Total
Number analyzed (Participants) | 463 | 441 | 904
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 463 | 441 | 904
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (.8) | 15.1 (.8) | 15.2 (.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 237 | 491
  Male | 209 | 204 | 413
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 283 | 314 | 597
  Native Hawaiian or other Pacific Islander | 3 | 1 | 4
  Native American or Alaska Native | 21 | 2 | 23
  Asian | 9 | 10 | 19
  Black or African American | 23 | 16 | 39
  Mixed race | 105 | 77 | 182
Region of Enrollment [Number; unit: participants]
  United States | 463 | 441 | 904

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent Students Eating the School Breakfast Per School
Description: Change in participation in the reimbursable school breakfast program will be evaluated from school provided objective participation data from baseline (SY1) to the end of one school year (SY2)
Time Frame: Change from baseline (SY1) in average school year school-level breakfast participation at the end of one school year (SY2).
Measure: Mean (Standard Deviation); unit: % School Breakfast Participation
Units Other Than Participants: Schools
Arm/Group | Intervention Arm | Comparison Arm
Number analyzed (Participants) | 463 | 441
Number analyzed (Schools) | 8 | 8
% School Breakfast Participation | 8.3 (9.8) | .9 (1.6)

2. Secondary Outcome: Change From Baseline in Body Mass Index
Description: Change from baseline to the end of one school year (SY2) in body mass index.
Time Frame: Change from baseline (SY1) in student body mass index at the end of one school year (SY2).
Population: The number of participants does not match that the the flow chart, and we were not able to to get post (SY2) BMI measures in all of the enrolled students.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Intervention Arm | Comparison Arm
Number analyzed (Participants) | 389 | 390
kg/m^2 | 1.0 (1.8) | .9 (1.6)

3. Secondary Outcome: Change From Baseline in Percent Body Fat
Description: Student percent body fat will be measured by trained research staff
Time Frame: Change from baseline in student body fat at the end of the school year (SY2)
Population: The number of participants does not match that the the flow chart, and we were not able to to get post (SY2) % body fat measures in all of the enrolled students.
Measure: Mean (Standard Deviation); unit: % Body Fat
Arm/Group | Intervention Arm | Comparison Arm
Number analyzed (Participants) | 389 | 390
% Body Fat | .1 (4.3) | -.2 (3.8)

4. Other Pre Specified Outcome: Change From Baseline in Healthy Eating Index Scores
Description: Change in the total Healthy Eating Index score from baseline to SY2. The Healthy Eating Index (HEI) score is a measure of diet quality. HEI scores can range from 0 to 100, with 0 representing the least overall healthy diet, and 100 representing the most overall healthy diet
Time Frame: Change from baseline in Healthy Eating Index at the end of the school year (SY2).
Population: The number of participants does not match that the the flow chart, and we were not able to to get post (SY2) HEI measures in all of the enrolled students.
Measure: Mean (Standard Deviation); unit: Healthy Eating Index Total Score
Arm/Group | Intervention Arm | Comparison Arm
Number analyzed (Participants) | 282 | 290
Healthy Eating Index Total Score | .6 (15.0) | -.3 (12.9)

5. Other Pre Specified Outcome: Social Support
Description: Change in social support from baseline to SY2. Assessment of social support for breakfast was measured by asking the students to consider a typical month and record how often the following people encouraged them to eat or continue to eat breakfast at school: (1) parent/guardian, (2) friend, (3) other kids at my school, (4) teacher, and (5) other school staff. A 4-point Likert-type scale (disagree to agree, 0-4) for each of the categories was used. The total scale summed the five categories. The scale ranged from 0-20, a higher score indicates more social support.
Time Frame: Change in perceived support from baseline at the end of the school year (SY2)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention Arm | Comparison Arm
Number analyzed (Participants) | 463 | 441
scores on a scale | .3 (3.4) | -.2 (3.9)

ADVERSE EVENTS:
Arm/Group | Intervention Arm | Comparison Arm
Serious Adverse Events (participants affected / at risk) | 0/463 | 0/441
Other Adverse Events (participants affected / at risk) | 0/463 | 0/441

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No